CLINICAL TRIAL: NCT01597505
Title: A Randomized, Double-Blinded, Active-Controlled Study of CB-183,315 in Patients With Clostridium Difficile Associated Diarrhea
Brief Title: Study of CB-183,315 in Participants With Clostridium Difficile Associated Diarrhea (MK-4261-005)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4261-005; LCD-CDAD-10-07 (Other: Cubist Study Number); MK-4261-005 (Other: Merck Protocol Number); 2012-000252-34 (EudraCT Number)
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Clostridium Difficile Infection
Keywords: CDAD; Clostridium difficile Associated Diarrhea; CDI; Clostridium difficile Infection; Diarrhea
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — CB-183,315; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surotomycin (Experimental): 250 mg Surotomycin over- encapsulated tablet administered orally, twice daily for a daily total dose of 500 mg; and Placebo over encapsulated tablet administered orally, twice daily for 10 days
  Interventions: Drug: Surotomycin; Drug: Placebo
- Vancomycin (Active Comparator): 125 mg Vancomycin over-encapsulated capsule administered orally, four times daily for a daily total dose of 500 mg, for 10 days
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Surotomycin — 250 mg Surotomycin over-encapsulated tablet administered orally, twice daily for a daily total dose of 500 mg, for 10 days
  Other Names: CB-183,315
  Arms: Surotomycin
Drug: Vancomycin — 125 mg Vancomycin over-encapsulated capsule administered orally, four times daily for a daily total dose of 500 mg, for 10 days
  Arms: Vancomycin
Drug: Placebo — Placebo for Surotomycin over-encapsulated tablet administered orally, twice daily for 10 days
  Arms: Surotomycin

SUMMARY:
606 participants with Clostridium Difficile Associated Diarrhea (CDAD) participated in this study and received either oral vancomycin or CB-183,315 (surotomycin) in a blinded fashion. Treatment lasted for 10 days and participants were followed up for at least 40 days and a maximum of 100 days. The purpose of this study was to evaluate how well surotomycin treats CDAD as compared to vancomycin.

ELIGIBILITY:
To be included in this study, participants must:

* Sign a consent form;
* Be >= 18 and < 90 years of age;
* Have diarrhea, at least 3 times during one day, or 200 mL or liquid stool if using a rectal device;
* Test positive for Clostridium difficile;
* If female, must not be pregnant or nursing and take appropriate measures to not get pregnant during the study.

Participants will not be allowed into the study if they:

* Have toxic megacolon and/or known small bowel ileus;
* Have received treatment with intravenous immune globulin (IVIG) within the past 30 days;
* Have received treatment with a fecal transplant within 7 days, and/or if the doctor anticipates to give the participant a fecal transplant during the study;
* Have received a certain amount of antibacterial therapy specific for current CDAD, unless it is not working;
* Have received an investigational vaccine against C. difficile;
* Have received an investigational product containing monoclonal antibodies against toxin A or B within 180 days;
* Had more than 2 episodes of CDAD within 90 days;
* Had major gastrointestinal (GI) surgery (i.e. significant bowel resection) within 3 months (this does not include appendectomy or cholecystectomy);
* Have history of prior inflammatory bowel disease: ulcerative colitis, Crohn's disease, or microscopic colitis;
* Are unable to discontinue loperamide, diphenoxylate/atropine, or cholestyramine during the duration of the study;
* Are unable to discontinue opiate treatment unless on a stable dose;
* Has known positive stool cultures for other enteropathogens including but not limited to Salmonella, Shigella, and Campylobacter;
* Had stool studies positive for pathogenic ova and/or parasites;
* Have an intolerance or hypersensitivity to daptomycin and/or vancomycin;
* Have life-threatening illness at the time of enrollment;
* Have poor concurrent medical risks that in the opinion of the Investigator the participant should not enroll;
* Have received an investigational drug or participated in any experimental procedure within 1 month;
* Have human immunodeficiency virus (HIV), a cluster of differentiation 4 (CD4) < 200 cells/mm3 within 6 months of start of study therapy;
* Anticipate that certain antibacterial therapy for a non-CDAD infection will be required for > 7 days;
* Are unable to discontinue Saccharomyces or similar probiotic;
* Are on a concurrent intensive induction chemotherapy, radiotherapy, or biologic treatment for active malignancy;
* Are unable to comply with the protocol requirements;
* Have any condition that, in the opinion of the Investigator, might interfere;
* Are not expected to live for less than 8 weeks.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2012-05-16 (Actual); Primary Completion 2015-03-20 (Actual); Study Completion 2015-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Boix V, Fedorak RN, Mullane KM, Pesant Y, Stoutenburgh U, Jin M, Adedoyin A, Chesnel L, Guris D, Larson KB, Murata Y. Primary Outcomes From a Phase 3, Randomized, Double-Blind, Active-Controlled Trial of Surotomycin in Subjects With Clostridium difficile Infection. Open Forum Infect Dis. 2017 Jan 19;4(1):ofw275. doi: 10.1093/ofid/ofw275. eCollection 2017 Winter. PMID 28480267
- [Derived] Cheknis A, Devaris D, Chesnel L, Dale SE, Nary J, Sambol SP, Citron DM, Goering RV, Johnson S. Characterization of Clostridioides difficile isolates recovered from two Phase 3 surotomycin treatment trials by restriction endonuclease analysis, PCR ribotyping and antimicrobial susceptibilities. J Antimicrob Chemother. 2020 Nov 1;75(11):3120-3125. doi: 10.1093/jac/dkaa297. PMID 32747931

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males and females aged 18 years or older with diarrhea at risk for Clostridium Difficile Associated Diarrhea (CDAD) were enrolled in this study
Groups:
- Surotomycin: 250 mg Surotomycin over encapsulated tablet administered orally, twice daily for a daily total dose of 500 mg; and Placebo over encapsulated tablet administered orally, twice daily for 10 days
Period: Overall Study
Arm/Group | Surotomycin | Vancomycin
Started | 308 (Randomized participants) | 298 (Randomized participants)
Treated | 305 (One participant was instead randomized to vancomycin) | 286
Completed | 264 | 265
Not Completed | 44 | 33
Not completed — Physician Decision | 5 | 0
Not completed — Adverse Event | 19 | 7
Not completed — Lost to Follow-up | 4 | 2
Not completed — Withdrawal by Subject | 10 | 18
Not completed — Other | 5 | 6
Not completed — Missing | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surotomycin | Vancomycin | Total
Number analyzed (Participants) | 308 | 298 | 606
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (17.5) | 61.8 (18.4) | 61.6 (17.9)
Age, Customized [Number; unit: Participants] — Number of participants <75 or >=75 years old at First Dose Population: Randomized participants with Confirmed CDAD
  Participants
    < 75 years old: number analyzed (Participants) | 290 | 280 | 570
    < 75 years old | 211 | 200 | 411
    >= 75 years old: number analyzed (Participants) | 290 | 280 | 570
    >= 75 years old | 79 | 80 | 159
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 175 | 360
  Male | 123 | 123 | 246
Previous episodes of CDAD [Number; unit: Participants] — Number of participants with previous episodes of CDAD Population: Randomized participants with Confirmed CDAD evaluated for previous episodes of CDAD
  Participants
    0 Previous Episodes: number analyzed (Participants) | 286 | 275 | 561
    0 Previous Episodes | 237 | 224 | 461
    >= 1 Previous Episodes: number analyzed (Participants) | 286 | 275 | 561
    >= 1 Previous Episodes | 49 | 51 | 100
BI/NAP1/027 Strain [Number; unit: Participants] — Number of participants with the BI/NAP1/027 Strain Population: Randomized participants with Confirmed CDAD evaluated for BI/NAP1/027 Strain
  Participants
    With BI/NAP1/027 Strain: number analyzed (Participants) | 255 | 246 | 501
    With BI/NAP1/027 Strain | 59 | 67 | 126
    Without BI/NAP1/027 Strain: number analyzed (Participants) | 255 | 246 | 501
    Without BI/NAP1/027 Strain | 196 | 179 | 375

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Percentage of Participants With a Clinical Outcome of Cure at the End of Treatment (EOT)
Description: A clinical outcome of cure at EOT was determined by resolution of diarrhea, defined as ≤ 2 loose stools per 24-hour period for at least 2 consecutive days and the lack of need for additional antibiotics to treat the current CDAD episode after completion of the study treatment period. Participants requiring a collection device were considered to have resolution of diarrhea when the volume of stool (over a 24-hour period) was decreased by 75% as compared to baseline or the participant was no longer passing liquid stool. The estimated adjusted percentage was a weighted average across all strata, constructed using Mehrotra-Railkar continuity-corrected minimum risk (MRc) stratum weights.
Time Frame: Up to 13 days
Population: The population analyzed is the Microbiological Modified Intent-To-Treat (mMITT) population consisting of all randomized participants who had a confirmed diagnosis of CDAD regardless of whether they received any amount of study drug, based on the treatment to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Surotomycin: 250 mg Surotomycin over encapsulated tablet administered orally, twice daily for a daily total dose of 500 mg for 10 days
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 290 | 280
Percentage of participants | 79.0 [73.9 to 83.2] | 83.6 [78.8 to 87.4]
Statistical Analysis 1: Comparison: Surotomycin vs Vancomycin; Difference in percentage of participants; Test type: Non-Inferiority — Surotomycin minus Vancomycin. For surotomycin to be non-inferior to vancomycin the lower bound of a 2-sided 95% CI for the difference between treatment groups had to be ≥ -10%; Difference in percentage of participants = -4.6, 95% CI 2-sided [-11.0 to 1.9] — The 95% confidence interval (CI) were stratified Wilson intervals for the treatment group percentages and a stratified Newcombe interval for the treatment difference, constructed using the MRc stratum weights

2. Secondary Outcome: Number of Participants With Clinical Response Over Time
Description: Clinical response over time as measured by those without treatment failure, recurrence, death, or lost to follow-up, measured as the number of participants without failure events (survivors) through the end of therapy (reported for Day 14) and from end of therapy to Day 40 (reported for Day 41).
Time Frame: Up to Day 41
Population: The mMITT population consisting of all randomized participants who had a confirmed diagnosis of CDAD regardless of whether they received any amount of study drug, based on the treatment to which they were randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 290 | 280
Participants
  Day 14 | 227 | 231
  Day 41 | 147 | 151
Statistical Analysis 1: Comparison: Surotomycin vs Vancomycin; Stratified log-rank test p-value; Test type: Superiority; p = 0.832, Log Rank — Log-rank test of equality of survival times, stratified by age group (< 75, >= 75 years) and number of CDAD episodes (0, >= 1). Significance cut-off = 0.05

3. Secondary Outcome: Adjusted Percentage of Participants With Sustained Clinical Response at the End of Study
Description: Sustained clinical response at the end of study was achieved by participants who had a clinical outcome of cure at the end of treatment (Days 40-50) and did not experience a recurrence of CDAD, did not die, were not lost to follow-up, and did not have end of study visit prior to Day 40. The estimated adjusted percentage was a weighted average across all strata, constructed using MRc stratum weights.
Time Frame: Up to Day 50
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 290 | 280
Percentage of participants | 60.6 [55.0 to 66.0] | 61.4 [55.9 to 66.8]
Statistical Analysis 1: Comparison: Surotomycin vs Vancomycin; Difference in percentage of participants; Test type: Superiority — Surotomycin - Vancomycin. For surotomycin to be considered superior to vancomycin the lower bound of the 2-sided 95% CI had to be > 0%; Difference in percentage of participants = -0.8, 95% CI 2-sided [-8.8 to 7.1] — The 95% CI was stratified Wilson intervals for group percentages and a stratified Newcombe interval for the difference, using the MRc stratum weights. Stratified by age group and number of CDAD episodes

4. Primary Outcome: Percentage of Participants With at Least One Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. AEs may be new events or may be pre-existing conditions that have become aggravated or have worsened in severity or frequency; or may be clinically significant changes from baseline in physical examination, laboratory tests, or other diagnostic investigation (e.g. laboratory results, x-ray findings).
Time Frame: Up to Day 50
Population: All randomized participants who received any amount of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 305 | 286
Percentage of participants | 48.5 | 55.2

5. Primary Outcome: Percentage of Participants With at Least One Serious Adverse Event (SAE)
Description: A SAE is any adverse experience occurring at any dose that results in any of the following outcomes: death; a life-threatening experience, referring to a situation in which the participant was at risk of death at the time of the event, requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability or incapacity; is a congenital anomaly or birth defect; or is considered to be an important medical event.
Time Frame: Up to Day 50
Population: All randomized participants who received any amount of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 305 | 286
Percentage of participants | 14.4 | 12.9

6. Primary Outcome: Percentage of Participants Who Discontinued Treatment Due to an AE
Description: as for outcome 4
Time Frame: Up to Day 13
Population: All randomized participants who received any amount of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 305 | 286
Percentage of participants | 5.6 | 2.8

7. Secondary Outcome: Adjusted Percentage of Participants With Sustained Clinical Response at Day 24
Description: Sustained clinical response at Day 24 was defined as participants who had a clinical outcome of cure at Day 24, who did not experience a recurrence of CDAD, did not die, were not lost to follow-up. Only the first failure event was counted per participant. The estimated adjusted percentage was a weighted average across all strata, constructed using MRc stratum weights.
Time Frame: Day 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 290 | 280
Percentage of participants | 66.6 [61.1 to 71.8] | 66.1 [60.5 to 71.3]
Statistical Analysis 1: Comparison: Surotomycin vs Vancomycin; Difference in percentage of participants; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Difference in percentage of participants = 0.6, 95% CI 2-sided [-7.2 to 8.3] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Adjusted Percentage of Participants With Recurrence of CDAD at End of Study
Description: Participants with recurrences were defined as those who were cured at the end of therapy and had a recurrence or were lost to follow-up, died or had a Day 40 -50 contact prior to Day 40. The estimated adjusted percentage was a weighted average across all strata, constructed using MRc stratum weights.
Time Frame: Up to Day 50
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 290 | 280
Percentage of participants | 17.7 [13.8 to 22.4] | 21.2 [16.9 to 26.1]
Statistical Analysis 1: Comparison: Surotomycin vs Vancomycin; Difference in percentage of participants; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Difference in percentage of participants = -3.5, 95% CI 2-sided [-10.0 to 3.0] — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Time to Resolution of Diarrhea
Description: Time to resolution of diarrhea with =< 2 unformed bowel movements (UBM) per 24-hour period was calculated as the date/time of last UBM minus the date/time of the first dose of study drug.
Time Frame: Up to Day 13
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 290 | 280
Days | 2.8 [2.2 to 3.3] | 3.0 [2.2 to 3.3]
Statistical Analysis 1: Comparison: Surotomycin vs Vancomycin; Stratified Log-Rank p-Value; Test type: Superiority — Surotomycin was superior to vancomycin if the p-value was less than 0.05; p = 0.431, Log Rank — [p-value comment as in outcome 2, analysis 1]

10. Secondary Outcome: Time to Reappearance of Diarrhea From End of Treatment to the End of Study
Description: Time to reappearance of diarrhea with >= 3 UBM per 24-hour period was calculated as the last date/time of study drug dose to the date/time of first reappearance of 3 or more UBMs among participants who were cured at end of treatment.
Time Frame: Up to Day 50
Population: The mMITT population consisting of all randomized participants who had a confirmed diagnosis of CDAD regardless of whether they received any amount of study drug, based on the treatment to which they were randomized; and were cured at end of treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 229 | 234
Days | NA [NA to NA] — The median value was not achieved | NA [NA to NA] — The median value was not achieved
Statistical Analysis 1: Comparison: Surotomycin vs Vancomycin; Stratified Log-Rank p-Value; Test type: Superiority — Surotomycin was superior to vancomycin if the p-value was less than 0.05; p = 0.011, Log Rank — [p-value comment as in outcome 2, analysis 1]

11. Secondary Outcome: Adjusted Percentage of Participants With a Clinical Response at the End of Treatment for Infections Deemed to be Caused by the C. Difficile BI/NAP1/027 Strain at Baseline
Description: Clinical response corresponded to a clinical outcome of cure at the end of treatment, and was achieved by participants with infections deemed to be caused by the C. difficile BI/NAP1/027 strain at baseline, who did not fail treatment, did not die, or were not lost to follow-up at the end of treatment. The estimated adjusted percentage was a weighted average across all strata, constructed using MRc stratum weights.
Time Frame: Up to Day 13
Population: Randomized participants who had a confirmed diagnosis of CDAD regardless of whether they received any amount of study drug, based on the treatment to which they were randomized; and with infections deemed to be caused by the C. difficile BI/NAP1/027 strain at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 59 | 67
Percentage of participants | 88.5 [75.8 to 92.4] | 86.3 [76.2 to 92.6]
Statistical Analysis 1: Comparison: Surotomycin vs Vancomycin; Difference in percentage of participants; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Difference in percentage of participants = 2.2, 95% CI 2-sided [-10.7 to 14.8] — Treatment group percentages were stratified by age group (< 75, ≥ 75) and number of previous CDAD episodes (0, ≥ 1). The 95% CIs were stratified Wilson intervals for the treatment group percentages

12. Secondary Outcome: Adjusted Percentage of Participants Per Protocol 1 Population With a Clinical Response at the End of Treatment
Description: Clinical response corresponded to a clinical outcome of cure at the end of treatment, and was achieved by participants who did not fail treatment, did not die, or were not lost to follow-up at the end of treatment. The estimated adjusted percentage was a weighted average across all strata, constructed using MRc stratum weights.
Time Frame: Up to Day 13
Population: The population analyzed is the Per Protocol 1 (PP1) population composed of participants from the mMITT population, according to the actual treatment they received; without any protocol deviations from enrollment through 2 days after end of treatment, which could affect the efficacy conclusions.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 252 | 243
Percentage of participants | 89.1 [84.5 to 92.2] | 91.5 [87.2 to 94.3]
Statistical Analysis 1: Comparison: Surotomycin vs Vancomycin; Difference in percentage of participants; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Difference in percentage of participants = -2.4, 95% CI 2-sided [-7.8 to 3.0] — Treatment group proportions were stratified by age group (< 75, ≥ 75) and number of previous CDAD episodes (0, ≥1). The 95% CIs were stratified Wilson intervals for the treatment group proportions

13. Secondary Outcome: Adjusted Percentage of Participants With a Sustained Clinical Response at the End of Study for Infections Deemed to be Caused by the C. Difficile BI/NAP1/027 Strain at Baseline
Description: Sustained clinical response at the end of study was achieved by participants with infections deemed to be caused by the C. difficile BI/NAP1/027 strain at baseline, who had a clinical outcome of cure at the end of treatment (Day 13) and did not experience a recurrence of CDAD, did not die, were not lost to follow-up, and did not have end of study visit prior to Day 40. The estimated adjusted percentage was a weighted average across all strata, constructed using MRc stratum weights.
Time Frame: Up to Day 50
Population: All randomized participants who had a confirmed diagnosis of CDAD regardless of whether they received any amount of study drug, based on the treatment to which they were randomized; and with infections deemed to be caused by the C. difficile BI/NAP1/027 strain at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 59 | 67
Percentage of participants | 66.1 [53.6 to 76.7] | 51.5 [40.5 to 63.1]
Statistical Analysis 1: Comparison: Surotomycin vs Vancomycin; Difference in percentage of participants; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Difference in percentage of participants = 14.6, 95% CI 2-sided [-2.7 to 30.7] — [estimate comment as in outcome 11, analysis 1]

14. Secondary Outcome: Adjusted Percentage of Participants From the Per Protocol 2 Population With a Sustained Clinical Response at the End of Study
Description: Sustained clinical response at the end of study was achieved by participants who had a clinical outcome of cure at the end of treatment (Days 40-50) and did not experience a recurrence of CDAD, did not die, were not lost to follow-up, and did not have end of study visit prior to Day 40. Only the first failure event per participant was counted. The estimated adjusted percentage was a weighted average across all strata, constructed using MRc stratum weights.
Time Frame: Up to Day 50
Population: The Per Protocol 2 (PP2) population composed of cures and failures from the PP1 population. Additionally, to be included in the PP2 population, PP1 participants who were cured at end of treatment must not have had any protocol deviations which could affect the assessment of recurrence and have had follow-up contact through at least Day 40.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Surotomycin | Vancomycin
Number analyzed (Participants) | 233 | 227
Percentage of participants | 70.8 [64.8 to 76.2] | 66.5 [60.6 to 72.2]
Statistical Analysis 1: Comparison: Surotomycin vs Vancomycin; Difference in percentage of participants; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Difference in percentage of participants = 4.3, 95% CI 2-sided [-4.2 to 12.7] — [estimate comment as in outcome 12, analysis 1]

ADVERSE EVENTS:
Time Frame: All AEs were collected up to Day 13; only SAEs and drug related AEs were collected thereafter 30 days after end of treatment (up to Day 50)
Description: All randomized participants who received any amount of study drug.
Groups:
- Surotomycin: 250 mg Surotomycin over-encapsulated tablet administered orally, twice daily for a daily total dose of 500 for 10 days
Arm/Group | Surotomycin | Vancomycin
All-Cause Mortality (participants affected / at risk) | 18/305 | 9/286
Serious Adverse Events (participants affected / at risk) | 44/305 | 37/286
Other Adverse Events (participants affected / at risk) | 38/305 | 38/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surotomycin (N=305) | Vancomycin (N=286)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (4) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Megacolon (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Sudden cardiac death (General disorders) | 2 (2) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Strongyloidiasis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tonic convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surotomycin (N=305) | Vancomycin (N=286)
Abdominal pain (Gastrointestinal disorders) | 16 (20) | 6 (6)
Nausea (Gastrointestinal disorders) | 20 (23) | 21 (21)
Headache (Nervous system disorders) | 12 (13) | 18 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No